CLINICAL TRIAL: NCT02819427
Title: Concomitant High-resolution Recording of Haemodynamic and Electrical Activities of Children With Typical or Atypical Absence Seizures: Near-infrared Spectroscopy (NIRS) Coupled to Electroencephalography (EEG)
Brief Title: Concomitant High-resolution Recording of Haemodynamic and Electrical Activities of Children With Typical or Atypical Absence Seizures
Acronym: Absence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2012_843_0025
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy
Keywords: Spectroscopy, Near-Infrared; Electroencephalography; children
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- epilepsy: children with absence epilepsy presenting either typical or atypical seizures
  Interventions: Device: Near Infra Red Spectroscopy (NIRS); Device: Electroencephalography (EEG)

INTERVENTIONS:
Device: Near Infra Red Spectroscopy (NIRS)
Device: Electroencephalography (EEG) — Electroencephalography (EEG) in a simultaneous High-Resolution (HR) recording.

SUMMARY:
This study, conducted in children with typical or atypical "absence" epilepsy, will consist of noninvasive recording of the metabolic activity of the brain concomitantly with electroencephalographic recording during seizures without the need for any additional examination. This examination will be performed by combining near-infrared spectroscopy (NIRS) optical imaging and Electroencephalography (EEG) in a simultaneous High-Resolution (HR) recording.

Surface electroencephalography (EEG) is a valuable tool to assess neuronal dysfunction from a functional point of view and is used in the routine follow-up of epileptic children. Optical imaging is a recent and promising medical imaging technique, which uses near-infrared light. This rapid, noninvasive and harmless quantitative technique can be easily used at the child's bedside or in the ward and provides metabolic information on brain functioning.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 14 years
* Featuring absence epilepsy with typical or atypical seizures characterized by the presence of spontaneous spike-wave flashes with standard EEG

Exclusion Criteria:

* All children with severe congenital malformation
* Any refusal of a parent or child
* Any child with a serious deterioration in the general condition and vital functions
* Any child with dermatitis of the face or scalp
* Children under 3 years old or over 14 years

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with absence epilepsy presenting either typical or atypical seizures
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
haemodynamic changes | Day 0
  haemodynamic changes by optical imaging, during the 4 interictal, preictal, ictal and postictal phases of absence seizures as defined by EEG analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice WALLOIS, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France